CLINICAL TRIAL: NCT00633412
Title: A Comparative Efficacy and Safety Study of Nexium Delayed-Release Capsules (40mg qd and 20mg qd) Versus Ranitidine 150mg Bid for the Healing of NSAID-Associated Gastric Ulcers When Daily NSAID Use is Continued in Subjects in the US Only
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH-NEN-0005; D9617C00005
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: NSAID Associated Gastric Ulcers
Keywords: NSAID; Nexium; esomeprazole; Gastric Ulcers
MeSH Terms: conditions — Stomach Ulcer | interventions — Esomeprazole; Ranitidine

ARMS (3):
- 1 (Experimental): 20mg Oral tablet daily
  Interventions: Drug: Esomeprazole
- 2 (Experimental): 40mg Oral tablet daily
  Interventions: Drug: Esomeprazole
- 3 (Active Comparator): 150mg oral twice daily
  Interventions: Drug: Ranitidine

INTERVENTIONS:
Drug: Esomeprazole — 20mg oral daily
  Other Names: Nexium
  Arms: 1
Drug: Ranitidine — 150mg oral twice daily
  Other Names: Zantac
  Arms: 3
Drug: Esomeprazole — 40mg oral tablet daily
  Other Names: Nexium
  Arms: 2

SUMMARY:
Nonsteroidal anti-inflammatory drugs (NSAIDS) are often associated with gastric ulcers. This study looks at the treatment of these gastric ulcers with one of the three following treatment groups for up to 8 weeks: esomeprazole 40 mg once daily; esomeprazole 20 mg once daily; or ranitidine 150 mg twice daily for subjects in the US only.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of a chronic condition (eg osteoarthritis or rheumatoid arthritis) that requires daily NSAID treatment for at least 2 months.
* A gastric ulcer >= 5mm in diameter, but no ulcer >25 mm at its greatest diameter, at the baseline endoscopy.
* Other key inclusion criteria, as specified in the protocol.

Exclusion Criteria:

* History of esophageal, gastric or duodenal surgery, except for simple closure of an ulcer.
* History of severe liver disease, including (but not limited to) cirrhosis and acute or chronic hepatitis.
* Many other conditions and criteria, as specified in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2001-02; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with no gastric ulcers after 8 weeks of treatment. | Esophagogastroduodenscopy (EGD) assessments at baseline, week 4, week 8, and efficacy evaluations at each visit including endoscopic evaluation for the presence of ulcers and erosions.

SECONDARY OUTCOMES:
The patient and investigator symptoms, defined as control of NSAID-associated GI symptoms up to 8 weeks of treatment with esomeprazole 40 mg vs ranitidine 150 mg bid and esomeprazole 20 mg qd versus ranitidine 150 mg bid in patients receiving daily N | Assessments at Week 0, Week 4 and Week 8
To look at any side effects of esomeprazole 40 mg vs ranitidine 150 mg bid and esomeprazole 20 mg qd versus ranitidine 150 mg bid in patients receiving daily NSAID therapy. | Assessments at Week 0, Week 4 and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca